CLINICAL TRIAL: NCT00725257
Title: Effect of a Low-Carbohydrate Mediterranean Diet or Low-Fat Diet in Newly-Diagnosed Type 2 Diabetic Patients
Brief Title: Dietary Control of Type 2 Diabetes: Low-Carbohydrate Mediterranean Diet Versus Low-Fat Diet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Department of Geriatrics and Metabolic Diseases
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DGMM/4/2004
Record Dates: First submitted 2008-07-28; First posted 2008-07-30 (Estimated); Last update posted 2008-07-30 (Estimated); Status verified 2008-07

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Diet, Mediterranean; Diet, Fat-Restricted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Low-carbohydrate, energy-restricted, Mediterranean-type diet
  Interventions: Other: Mediterranean diet
- 2 (Active Comparator): Low-fat diet
  Interventions: Other: Low-fat diet

INTERVENTIONS:
Other: Mediterranean diet — The recommended composition of the dietary regimen was as follows: Carbohydrate 40 to 50%, protein 15 to 20%; fat 30 to 40%; saturated fat less than 10%.
  Arms: 1
Other: Low-fat diet — The recommended composition of the dietary regimen was as follows: Fat less than 30%; carbohydrate 50 to 60%, protein 15 to 20%; saturated fat less than 10%.
  Arms: 2

SUMMARY:
The major environmental factors that increase the risk of type 2 diabetes, presumably in the setting of genetic risk, are overnutrition and a sedentary lifestyle, with consequent overweight and obesity. The high rate of weight regain has limited the role of lifestyle interventions as an effective means of controlling glycemia long term. The aims of the present study were: 1) To compare the effectiveness and safety of two nutritional protocols - namely low-carbohydrate Mediterranean diet or low-fat diet - in newly-diagnosed, drug-naive overweight patients with type 2 diabetes mellitus. The primary aim of the study was the effect on hemoglobin A1c levels; secondary aims were time to introduction of the first hypoglycemic agent, prevalence of the metabolic syndrome, percentage of patients meeting ADA goals for risk factors (HbA1c, blood pressure, LDL-cholesterol, percentage of patients with HbA1c < 7%.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus (ADA criteria)
* BMI (body mass index) > 25 kg/M2
* Hemoglobin A1c (HbA1c) < 11%; Blood pressure < 160 (systolic) and 100 (diastolic) mm Hg
* Triglyceride levels < 500 mg/dl.

Exclusion Criteria:

* Pregnancy or breast-feeding
* Previous use of insulin or oral antidiabetic drugs
* Investigational drug within the previous 3 months
* Use of agents affecting glycemic control (systemic steroids and weight loss drugs)
* Patients with history of alcohol or illicit drug abuse
* Patients with liver enzymes higher than three times the upper limit of normal
* Serum creatinine > 1.4 mg/dl.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2004-06; Primary Completion 2007-09 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1c | Every sixth month

SECONDARY OUTCOMES:
Time to introduction of an oral hypoglycemic agent | Every year

CONTACTS AND LOCATIONS:
Overall Officials: Dario Giugliano, MD,PhD, Principal Investigator — Department of Geriatrics and Metabolic Diseases
Locations (1):
- Department of Geriatrics and Metabolic Diseases, Naples, Italy

REFERENCES:
- [Background] Shai I, Schwarzfuchs D, Henkin Y, Shahar DR, Witkow S, Greenberg I, Golan R, Fraser D, Bolotin A, Vardi H, Tangi-Rozental O, Zuk-Ramot R, Sarusi B, Brickner D, Schwartz Z, Sheiner E, Marko R, Katorza E, Thiery J, Fiedler GM, Bluher M, Stumvoll M, Stampfer MJ; Dietary Intervention Randomized Controlled Trial (DIRECT) Group. Weight loss with a low-carbohydrate, Mediterranean, or low-fat diet. N Engl J Med. 2008 Jul 17;359(3):229-41. doi: 10.1056/NEJMoa0708681. PMID 18635428
- [Background] Esposito K, Ciotola M, Giugliano D. Low-carbohydrate diet and coronary heart disease in women. N Engl J Med. 2007 Feb 15;356(7):750; author reply 750-2. doi: 10.1056/NEJMc063464. No abstract available. PMID 17301311
- [Derived] Maiorino MI, Bellastella G, Petrizzo M, Gicchino M, Caputo M, Giugliano D, Esposito K. Effect of a Mediterranean diet on endothelial progenitor cells and carotid intima-media thickness in type 2 diabetes: Follow-up of a randomized trial. Eur J Prev Cardiol. 2017 Mar;24(4):399-408. doi: 10.1177/2047487316676133. Epub 2016 Oct 27. PMID 27798369
- [Derived] Maiorino MI, Bellastella G, Caputo M, Castaldo F, Improta MR, Giugliano D, Esposito K. Effects of Mediterranean diet on sexual function in people with newly diagnosed type 2 diabetes: The MEDITA trial. J Diabetes Complications. 2016 Nov-Dec;30(8):1519-1524. doi: 10.1016/j.jdiacomp.2016.08.007. Epub 2016 Aug 12. PMID 27614727
- [Derived] Maiorino MI, Bellastella G, Chiodini P, Romano O, Scappaticcio L, Giugliano D, Esposito K. Primary Prevention of Sexual Dysfunction With Mediterranean Diet in Type 2 Diabetes: The MEDITA Randomized Trial. Diabetes Care. 2016 Sep;39(9):e143-4. doi: 10.2337/dc16-0910. Epub 2016 Jun 28. No abstract available. PMID 27352954
- [Derived] Maiorino MI, Bellastella G, Petrizzo M, Scappaticcio L, Giugliano D, Esposito K. Anti-inflammatory Effect of Mediterranean Diet in Type 2 Diabetes Is Durable: 8-Year Follow-up of a Controlled Trial. Diabetes Care. 2016 Mar;39(3):e44-5. doi: 10.2337/dc15-2356. Epub 2016 Jan 6. No abstract available. PMID 26740638
- [Derived] Esposito K, Maiorino MI, Petrizzo M, Bellastella G, Giugliano D. The effects of a Mediterranean diet on the need for diabetes drugs and remission of newly diagnosed type 2 diabetes: follow-up of a randomized trial. Diabetes Care. 2014 Jul;37(7):1824-30. doi: 10.2337/dc13-2899. Epub 2014 Apr 10. PMID 24722497